CLINICAL TRIAL: NCT07272928
Title: Comparison of the Resection Site Order in Simultaneous Approach of Colorectal Liver Metastasis. An International Multicentric Retrospective Trial.
Brief Title: Comparison of the Resection Site Order in Simultaneous Approach of Colorectal Liver Metastasis
Acronym: CORSICO
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.ChirGen.24.06
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Liver Metastasis
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Data collection — Data collection to assess whether the order of resection of the site in a simultaneous approach (liver first vs. colon first) in colorectal cancer with liver metastases affects overall postoperative morbidity.

SUMMARY:
Colorectal cancer frequently presents with liver metastases, and complete removal of both primary and liver tumors can significantly improve survival. Simultaneous resection (SA) of the colon and liver is increasingly used and is considered safe when minor liver resections are performed, offering advantages such as shorter hospitalization, fewer complications, and faster chemotherapy initiation.

However, the best sequence of resection, liver-first or colon-first, remains uncertain, as each has potential benefits and drawbacks, particularly regarding anastomotic healing. Minimally invasive approaches to SA show similar outcomes to open surgery, though limited data suggest that resection order may affect blood loss.

DETAILED DESCRIPTION:
Colorectal cancer is the third most common cancer worldwide, and 15-25% of patients present with liver metastases at diagnosis. Complete resection of both the primary tumor and liver metastases can yield survival rates up to 47.9%. Simultaneous resection (SA) of the colon and liver is a potential option for patients with synchronous metastases, though traditionally considered high-risk, especially when major hepatectomies are involved.

Recent studies show that SA is safe when minor hepatectomies are paired with standard colon resections and may offer advantages such as reduced hospital stay, lower costs, fewer complications, and faster initiation of chemotherapy.

The optimal sequence of resection in SA remains unclear. Liver-first procedures may preserve sterility and address the prognostically significant lesion first but could impair bowel anastomosis healing.

Minimally invasive surgery (MIS), including laparoscopic and robotic approaches, is increasingly used for SA and appears comparable to open surgery in terms of morbidity, mortality, and oncologic outcomes. Early data on MIS suggest that resection order may influence intraoperative blood loss, but findings remain inconsistent and require further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with colorectal cancer with synchronous liver metastases during the reference period, who underwent simultaneous resection.

Exclusion Criteria:

* Simultaneous emergency resection due to symptoms of the primary tumor.
* Presence of extrahepatic metastatic disease confirmed at the time of resection or diagnosis.
* High surgical risk defined as an ASA risk score greater than 3.
* At least 10 cases performed by the invited center during the study period.
* Incomplete data or follow-up of less than 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing simultaneous treatment of colorectal cancer and liver metastases using open, laparoscopic, and robotic surgery between 2015 and 2023 in participating centers
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
Difference in overall morbidity rates | Through study completion, an average of 1 year
  Measurement of the difference in overall morbidity rates between both approaches (liver first vs. colon first) in colorectal cancer with liver metastasis influences postoperative

SECONDARY OUTCOMES:
Mortality | Through study completion, an average of 1 year
  Evaluation of the postoperative mortality for both approaches, (liver first vs. colon first), when performed via laparoscopic or robotic surgery
Overall survival | Through study completion, an average of 1 year
  Compare the overall survival of patients with a diagnosis of colorectal cancer between both approaches (liver first vs. colon first), when performed via laparoscopic or robotic surgery
Disease-free survival | Through study completion, an average of 1 year
  Compare the disease-free survival of patients with a diagnosis of colorectal cancer between both approaches (liver first vs. colon first), when performed via laparoscopic or robotic surgery
Recurrence sites | Through study completion, an average of 1 year
  Compare the recurrence sites in patients with a diagnosis of colorectal cancer between both approaches (liver first vs. colon first), when performed via laparoscopic or robotic surgery
Morbidity | Through study completion, an average of 1 year
  Compare the morbidity in patients with a diagnosis of colorectal cancer between both approaches (liver first vs. colon first), when performed via laparoscopic or robotic surgery

CONTACTS AND LOCATIONS:
Locations (1):
- SC Chirurgia Generale, Alessandria, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No